CLINICAL TRIAL: NCT00474227
Title: Proper Nutrition, Physical Exercise and Appropriate Weight in Individuals With Long Term Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lev-Hasharon Mental Healtlh Center (Other Government)
Responsible Party: Gloria Ilievici, MD, Lev Hasharon Mental Health Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LH33/2007.CTIL
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-05

CONDITIONS: Obesity
Keywords: obesity; weight gain; schizophrenia; schizoaffective disorder; antipsychotic induced weight gain
MeSH Terms: conditions — Obesity; Weight Gain; Schizophrenia; Psychotic Disorders | interventions — Psychotherapy, Group; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): behavioral intervention, group therapy including nutritional guidance and physical exercise
  Interventions: Behavioral: group therapy, physical exercise, nutrition lectures
- B (No Intervention): comparison group, one time explanation of importance of proper nutrition. This group receives no group therapy or organized exercise sessions or nutritional guidance. They are wait listed for this program.

INTERVENTIONS:
Behavioral: group therapy, physical exercise, nutrition lectures — weekly group therapy, physical exercize, nutrition guidance
  Arms: A

SUMMARY:
Based on previous findings that mentally ill inpatients are interested in losing treatment associate weight gain and are capable of adhering to a weight reduction program, this study will investigate the effects of participation in nutrition intervention, physical exercise and will monitor measurement of metabolic profiles (cholesterol, triglycerides and glucose). Hypothesis: participants will reduce weight, maintain weight loss and experience reduction in metabolic values and will experience improved quality of life.

DETAILED DESCRIPTION:
Study sample: 50 chronic psychiatric inpatients with DSM_IV diagnosis of schizophrenia or schizoaffective disorder, aged 18 or older. Exclusion criteria - pregnancy, severe physical illness, refusal to participate.

Study instruments: Q-LES-Q-18 (quality of life): Positive and Negative Syndrome Scale; Laboratory test- glucose levels, metabolic profiles (cholesterol, triglycerides). Measurements: Weight, BMI, pulse Intervention: Weekly group therapy, lectures on nutrition, physical exercise Duration of study: 3 months

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* Men or women
* Schizophrenia or schizoaffective disorder
* BMI greater than 26
* Agreement to participate and capacity to provide written informed consent

Exclusion Criteria:

* Pregnancy
* Severe physical illness
* Refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
weight reduction | three months

SECONDARY OUTCOMES:
improved metabolic profile | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Ilievici, MD, Principal Investigator — Lev HaSharon Mental Health Center; Yuval Melamed, MD, MHA, Study Director — Lev HaSharon Mental Health Center
Locations (1):
- Lev Hasharon Mental Health Center, Netanya, Israel

REFERENCES:
- See also: website of location of study — http://www.lev-hasharon.co.il